CLINICAL TRIAL: NCT06901700
Title: Effects of Home-based Lower Extremity Muscle Power Training on Functional Muscle and Balance Performance in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU114046AF
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-03

CONDITIONS: Older Adults
Keywords: Power training; Home-based training; Muscle performance; Balance; Older adults
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Health education
  Interventions: Other: control group
- Experimental group (Experimental): Total 40~60 minutes, 3 sessions per week in alternate day for 8 weeks, total 24 sessions
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — Total 40~60 minutes, 3 sessions per week in alternate day for 8 weeks, total 24 sessions 5 min warm up and 5 min cool down Power training (using body weight as resistance): hip flexor, hip extensor, hip adductor, hip abductor, knee flexor, ankle plantarflexor, hip external rotator, hip internal rotator, knee extensor, ankle dorsiflexor, ankle invertor, ankle evertor
  Arms: Experimental group
Other: control group — Health education
  Arms: Control group

SUMMARY:
Background: Muscle power, defined as the rate at which muscular force is generated to produce movement, declines more rapidly with age than muscle strength. The decline in lower extremity muscle power is associated with reduced functional independence, impaired mobility, and an increased risk of falls among older adults. While power training has been shown to improve muscle power, balance, and functional abilities, the feasibility and effectiveness of home-based interventions have not been thoroughly investigated.

Purpose: The aim of this study is to investigate the effects of home-based lower extremity muscle power training program on functional muscle and balance performance in older adults.

Methods: This is a single-blind, randomized controlled trial. Forty community-dwelling older adults will be recruited and randomly assigned to the experimental group (n=20) and control group (n=20). Participants in the experimental group will complete 24 sessions of home-based lower extremity muscle power training targeting the lower limb muscle groups in 8 weeks. The training intensity will be progressively adjusted according to participants' performance. Participants in the control group will maintain their daily activities. In addition, both groups will receive health education. Primary outcomes include functional muscle power measured by the Four-Step Stair Climb Power Test, functional muscle strength measured by Five Times Sit-to-Stand Test, and the functional balance performance measured by the Mini-BESTest, and Timed Up and Go Test. The fall confidence, as the secondary outcome, will be measured by Falls Efficacy Scale International.

Statistical analysis: The SPSS® version 29 will be used for statistical analysis. Independent-t-test or chi-square test will be conducted to compare the baseline demographic characteristics between groups. Two-way repeated measure ANOVA will be used to compare the differences between groups and times, post-hoc analyses will be performed using Tukey's test. The significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 65~80 years old community-dwelling adults
* MMSE≥24
* Use smart phone routinely

Exclusion Criteria:

* Recent (<1 year) musculoskeletal injury or disability in the lower limbs
* Unstable cardiovascular, neurological disease, or metabolic disease interfering with participating in the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Functional muscle performance-muscle power | From baseline to the end of treatment at 8 weeks
  The Four-Step Stair Climb Power Test is used for measurement, where participants rapidly ascend four steps while the required time is recorded. This test is designed to assess lower limb muscle power.
Functional muscle performance-muscle strength | From baseline to the end of treatment at 8 weeks
  The 5 Times Sit-to-Stand Test is used for measurement, where participants quickly and continuously perform five sit-to-stand movements while the required time is recorded. This test is designed to assess lower limb muscle strength.
Balance | From baseline to the end of treatment at 8 weeks
  The Mini-BESTest (Balance Evaluation Systems Test) is used for measurement. This test includes anticipatory control, reactive postural control, sensory orientation, and dynamic gait, allowing for the assessment of balance abilities related to postural control.
Timed Up and Go Test | From baseline to the end of treatment at 8 weeks
  The Timed Up and Go (TUG) Test is conducted at both a normal and fast pace to assess the balance and mobility of community-dwelling older adults in functional activities.

SECONDARY OUTCOMES:
Fall confidence | From baseline to the end of treatment at 8 weeks
  The Falls Efficacy Scale International (FES-I) is used for assessment. This scale evaluates the level of confidence in not falling while performing activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No